CLINICAL TRIAL: NCT05392192
Title: A Randomized, Double-Blind, Placebo-Controlled, Two-Period Crossover, Phase 2 Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of ADX-629 Administered Orally to Subjects With Chronic Cough
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy in Subjects With Chronic Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-629-CC-001
Record Dates: First submitted 2022-05-05; First posted 2022-05-26 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2022-07

CONDITIONS: Chronic Cough
Keywords: refractory cough; cough hypersensitivity; ADX-629; unexplained cough; reactive aldehyde species; crossover; inflammation
MeSH Terms: conditions — Chronic Cough; Cough; Inflammation | interventions — ADX-629

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADX-629 (Experimental): Subjects will be randomized to receive ADX-629 300mg tablets administered orally twice a day for 14 days.
  Interventions: Drug: ADX-629
- Placebo (Placebo Comparator): Subjects will be randomized to receive matching placebo tablets administered orally twice a day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX-629 — Subjects will be randomized to receive both ADX-629 and placebo in one of two treatment sequences: One group of subjects will receive ADX-629 during the 1st treatment period and matching placebo during the 2nd Treatment while subjects the other sequence/group will receive the matching placebo in the 1st treatment period and ADX-629 in the 2nd treatment period.
  Arms: ADX-629
Drug: Placebo — Subjects will be randomized to receive both ADX-629 and placebo in one of two treatment sequences: One group of subjects will receive ADX-629 during the 1st treatment period and matching placebo during the 2nd Treatment while subjects the other sequence/group will receive the matching placebo in the 1st treatment period and ADX-629 in the 2nd treatment period.
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Two-Period Crossover, Phase 2 Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of ADX-629 Administered Orally to Subjects with Chronic Cough

DETAILED DESCRIPTION:
A Phase 2, multicenter, randomized, double-blind, placebo controlled, two-period crossover trial to evaluate the safety, tolerability, and efficacy of ADX-629 (300 mg) administered orally, twice-a-day to eligible participants with refractory or unexplained chronic cough. Patients who are interested in participating will be provided detailed information about the study including description of study assessments/procedures, possible side-effects, alternative treatments, and potential benefits.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 to ≤80 years of age
* History of refractory or unexplained chronic cough
* Historical Chest radiograph or CT scan that does not demonstrate any abnormality considered to be significantly contributing to chronic cough
* Not pregnant, breastfeeding, or lactating and agree to use a highly effective method of acceptable contraceptive for the trial duration, if applicable
* Agree to discontinue antitussive medications for the trial duration

Exclusion Criteria:

* Current smoker (including cannabis products) or previous smoker having recently given up smoking or has a history of smoking of >20 pack-years
* History of significant cardiovascular disease or any clinically significant abnormalities in rhythm or conduction
* History or presence of significant hepatic disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of any malignancy within 5 years of screening except for basal cell or squamous cell in situ skin carcinomas or carcinoma in situ of the cervix that has been treated with no evidence of recurrence.
* Recent history of drug or alcohol abuse or a positive urine drug test at screening
* Positive serology test for Hepatitis B virus (HBV), Hepatitis C virus (HCV), or HIV-1 and HIV-2
* Currently taking an angiotensin converting enzyme inhibitor (ACEI) or has used an ACEI within 3 months of Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Allergy Associates Medical Group, Inc., San Diego, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - Cano Research - Hollywood, Hollywood, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - Florida Pulmonary Research Institute LLC, Winter Park, Florida
  - ClinCept, Columbus, Georgia
  - Mayo Clinic Pulmonary Clinic Research Unit, Rochester, Minnesota
  - Mount Sinai, New York, New York
  - Charlotte Lung & Health/American Health Research, Charlotte, North Carolina
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Vital Prospects Clinical Research, Tulsa, Oklahoma
  - Northwest Research Center, Portland, Oregon
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Pharmaceutical Research and Consulting Inc., Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty-one subjects were randomized in a crossover design.
Groups:
- ADX-629 First, Then Placebo: ADX-629 300mg (milligrams) administered orally twice daily (BID) for two weeks, followed by a two-week washout, then placebo administered orally BID for two weeks.
- Placebo First, Then ADX-629: Placebo administered orally BID for two weeks, followed by a two-week washout, then ADX-629 300mg administered orally BID for two weeks.
Period: Overall Study
Arm/Group | ADX-629 First, Then Placebo | Placebo First, Then ADX-629
Started | 26 | 25
Completed | 26 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- ADX-629 First, Then Placebo: ADX-629 300mg administered orally BID for two weeks, followed by a two-week washout, then placebo administered orally BID for two weeks.
- Total: Total of all reporting groups
Arm/Group | ADX-629 First, Then Placebo | Placebo First, Then ADX-629 | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (9.5) | 65.2 (7.1) | 65.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 23 | 24 | 47
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.4 (9.5) | 28.4 (4.7) | 28.9 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events
Description: Safety was assessed through serious adverse event collection.
Time Frame: The safety assessment period was Day 1 - Day 14 for each treatment period.
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- ADX-629: ADX-629 300mg administered orally BID for 14 days.
- Placebo: Placebo administered orally BID for 14 days.
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 47 | 51
Participants | 0 | 0

2. Secondary Outcome: Change From Baseline in Awake Cough Frequency Per Hour With Prior Treatment as a Factor
Description: Change from baseline in cough count was assessed while subjects were awake using a cough monitor with a digital recording device. The number of coughs is proportional to disease severity. Estimates were obtained using mixed model repeated measures (MMRM) analysis with treatment and prior treatment (none for Period 1; Period 1 treatment for Period 2) as fixed effects, and period-specific baseline as a covariate.
Time Frame: The efficacy assessment period was Day 14 for each treatment period. Baseline was Day 1 prior to dosing for each treatment period.
Population: Intent-to-treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: coughs per hour
Groups:
- ADX-629: ADX-629 300mg administered orally BID for two weeks
- Placebo: Placebo administered orally BID for two weeks
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 47 | 51
coughs per hour | -7.06 [-14.44 to 0.31] | 7.68 [0.78 to 14.58]

3. Secondary Outcome: Change From Baseline in 24-hour Cough Frequency Per Hour With Prior Treatment as a Factor
Description: Change from baseline in cough count was assessed for twenty-four hours using a cough monitor with a digital recording device. Number of coughs is associated with disease severity. Estimates were obtained using MMRM analysis with treatment and prior treatment (none for Period 1; Period 1 treatment for Period 2) as fixed effects, and period-specific baseline as a covariate.
Time Frame: as for outcome 2
Population: Intent-to-treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: coughs per hour
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 47 | 51
coughs per hour | -5.57 [-10.20 to -0.93] | 6.39 [2.04 to 10.75]

4. Secondary Outcome: Change From Baseline in Awake Cough Frequency Per Hour for Period 1
Description: Change from baseline in cough count in Period 1 was assessed while subjects were awake using a cough monitor with a digital recording device. The number of coughs is proportional to disease severity. Estimates were obtained using MMRM analysis with treatment as fixed effect, and Period 1-specific baseline as a covariate.
Time Frame: The efficacy assessment period was Day 14. Baseline was Day 1 for Period 1.
Population: Intent-to-treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: coughs per hour
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 24 | 25
coughs per hour | -11.51 [-19.78 to -3.24] | 2.45 [-5.65 to 10.56]

5. Secondary Outcome: Change From Baseline in 24-hour Cough Frequency Per Hour for Period 1
Description: Change from baseline in cough count in Period 1 was assessed for twenty-four hours using a cough monitor with a digital recording device. The number of coughs is proportional to disease severity. Estimates were obtained using MMRM analysis with treatment as fixed effect, and Period 1-specific baseline as a covariate.
Time Frame: The efficacy assessment period was Day 14. Baseline was Day 1 for Period 1.
Population: Intent-to-treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: coughs per hour
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 24 | 25
coughs per hour | -9.39 [-14.80 to -3.99] | 2.02 [-3.27 to 7.32]

ADVERSE EVENTS:
Time Frame: Fourteen days for each intervention
Arm/Group | ADX-629 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 3/51 | 0/51
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADX-629 (N=51) | Placebo (N=51)
Headache (Nervous system disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT05392192/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT05392192/SAP_001.pdf